CLINICAL TRIAL: NCT05064748
Title: A Multi-center, Open-Label, Extension Study to Evaluate the Safety and Efficacy of Benvitimod Cream in the Treatment of Mild to Moderate Psoriasis in Adults
Brief Title: Phase IV Clinical Study of Benvitimod Cream in the Treatment of Mild to Moderate Psoriasis in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Zhonghao Pharmaceutical (Unknown)
Responsible Party: Principal Investigator, Zhang jianzhong, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ202105BWMD
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis
Keywords: Benvitimod Cream; Psoriasis; Topical Treatment
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental)
  Interventions: Drug: Benvitimod

INTERVENTIONS:
Drug: Benvitimod — Benvitimod cream, 1%, applied twice daily for 12 weeks after enrolment.

SUMMARY:
This is a multi-center, prospective post-approval clinical Phase IV study to evaluate the safety and efficacy of Benvitimod cream, 1% twice daily for the treatment of mild to moderate stable psoriasis vulgaris in adults. Approximately 2000 adult participants with mild to moderate stable psoriasis vulgaris will be enrolled and they will use the Benvitimod cream at the skin with psoriasis for 12 weeks.

DETAILED DESCRIPTION:
This is a multi-center, prospective post-approval clinical Phase IV study to evaluate the safety and efficacy of Benvitimod cream, 1% twice daily for the treatment of mild to moderate stable psoriasis vulgaris in adults. Approximately 2000 adult participants with mild to moderate stable psoriasis vulgaris will be enrolled and they will apply the Benvitimod cream on the skin with plaque psoriasis for maximum 12 weeks. All participants will complete follow-up visits at 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks and continuing up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ages at least 18 years.
* The participant with diagnosis of mild to moderate stable psoriasis vulgaris.
* BSA involvement <10%.
* Capable of giving written informed consent.

Exclusion Criteria:

* Planned Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation during the study period.
* Known allergies to the active ingredient or excipients of the drug.
* Pregnant females, lactating females.
* The patients who were considered unsuitable to participate in the study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) from Baseline to Week 12 | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Percentage decline in Physician Global Assessment (PGA) score at Week 12 | Week 12
  The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis at a given timepoint. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, scaling, and plaque thickness/elevation as guidelines. Higher PGA scores represent more severe disease.

SECONDARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) from Baseline to Week 8 | Week 8
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥90% improvement in Psoriasis Area and Severity Index (PASI) score from Baseline to Week 8 | Week 8
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥75% improvement in Psoriasis Area and Severity Index (PASI) score from Baseline to Week 8 | Week 8
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥50% improvement in Psoriasis Area and Severity Index (PASI) score from Baseline to Week 8 | Week 8
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Change in percent of total body surface area (%BSA) affected from Baseline to Week 8 | Week 8
  The assessment of %BSA affected is an estimate of the percentage of total involved skin with psoriasis. For the purpose of clinical estimation, the total palmar surface of the participant's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by psoriasis will be evaluated (from 0% to 100%). %BSA is a static assessment made without reference to previous scores.
Proportion of participants with ≥90% improvement in Psoriasis Area and Severity Index (PASI) score from Baseline to Week 12 | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥75% improvement in Psoriasis Area and Severity Index (PASI) score from Baseline to Week 12 | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Proportion of participants with ≥50% improvement in Psoriasis Area and Severity Index (PASI) score from Baseline to Week 12 | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Change in percent of total body surface area (%BSA) affected from Baseline to Week 12 | Week 12
  The assessment of %BSA affected is an estimate of the percentage of total involved skin with psoriasis. For the purpose of clinical estimation, the total palmar surface of the participant's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by psoriasis will be evaluated (from 0% to 100%). %BSA is a static assessment made without reference to previous scores.
Change of Psoriasis Area and Severity Index (PASI) score over time from Baseline to Week 12. | Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
The Dermatology Life Quality Index (DLQI) total and individual dimension scores. | Week 16
  The DLQI is a simple dermatology-specific 10-question validated questionnaire to assess the impact of the disease on a participant's quality of life. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
European Questionnaires Five Dimensions Five Levels (EQ-5D-5L) scores. | Week 16
  EQ-5D-5L is a standardized instrument for measuring generic health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided